CLINICAL TRIAL: NCT03137914
Title: Clinical Study for the Evaluation of the Safety and Effectiveness of Autologous Chondrocytes Transplantation for the Treatment of Condylar Resorption Associated With Dentofacial Deformities
Brief Title: Nasal Septum Autologous Chondrocytes Transplantation for Condylar Resorption After Orthognathic Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Faculdade de Medicina de Petrópolis Faculdade Arthur Sá Earp Neto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U111111946997
Record Dates: First submitted 2017-04-25; First posted 2017-05-03 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Temporomandibular Joint Disorders
Keywords: orthognathic surgery; TMJ; osteoarthritis
MeSH Terms: conditions — Temporomandibular Joint Disorders; Osteoarthritis | interventions — Orthognathic Surgery

STUDY DESIGN:
Intervention Model Description: Single Group Assignment The clinical study model adopted is a single experimental group. Ten participants with dentofacial deformities related to severe degenerative TMJ changes, who are candidates for orthognathic surgery to repair these deformities, will be evaluated, who will be submitted to treatment with nasal septum autologous chondrocytes transplantation. There will be no evaluation of the control group in this study, as it is a case report. Injection of the experimental treatment will be done through an ultrasound-guided arthrocentesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- autologous chondrocyte transplantation (Experimental): Autologous transplant of chondrocytes diluted in hyaluronic acid after orthognathic surgery. The transplantation will be performed through an intra-articular injection into the TMJ (arthrocentesis). Hyaluronic acid is used only as a soluble medium to dilute the chondrocytes, so it is not considered as another experimental group, or as part of interest in this investigation.
  Interventions: Biological: Autologous chondrocyte transplantation; Procedure: orthognathic surgery

INTERVENTIONS:
Biological: Autologous chondrocyte transplantation — intraarticular injection into the TMJ (arthrocentesis) of autologous chondrocytes diluted in hyaluronic acid
Procedure: orthognathic surgery — Orthognathic surgery for correction of dentofacial deformity, performed before the cellular transplantation

SUMMARY:
This clinical study has as main objective to evaluate if the Nasal Septum Autologous Chondrocytes Transplantation for Condylar Resorption is safe and effective in the treatment of degenerative lesions of temporomandibular joint (TMJ). It is a case series, in which 10 participants with diagnosis of condylar reabsorption of TMJ will be selected, with orthognathic surgery indicated. Orthognathic surgery is conventionally indicated for patients with condylar resorption to correct dentofacial deformity and, therefore, will not be performed only in function of this clinical study. The selected participants will be submitted to nasal cartilage biopsy, for isolation and preparation of the chondrocytes. The only experimental group to be evaluated will be the group treated with autologous chondrocytes diluted in hyaluronic acid. The experimental treatment will be performed 15 days after orthognathic surgery, and will be injected through arthrocentesis. Clinical follow- up will be performed in the following periods: 7 and 15 days and 1, 3, 6 and 12 months after treatment. During the consultations, participants will also be evaluated for the intensity and severity of the pain experienced, as well as the disability related to it, through the same system used for the diagnostic classification (RDC / TMD). Imaging of the TMJ will be performed before, 6 and 12 months after the injection of the experimental treatment for bone and cartilaginous joint tissue analysis. Autologous chondrocyte implantation is expected to promote the regeneration of TMJ cartilage tissue safely and effectively.

DETAILED DESCRIPTION:
The only experimental group to be evaluated will be the group treated with autologous chondrocytes diluted in hyaluronic acid, to be included in groups of 2, 4 and 4 participants. Only two participants will initially be included. If these two treated participants do not present adverse effects in 3 months, we will start a second stage with 4 participants. Again we will analyze the group over 3 months and if there are no problems we will include the 4 final participants, totaling the 10 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of dentofacial deformities related to osteoarthritis of TMJ;
2. must have surgical indication.

Exclusion Criteria:

1. pregnant or breastfeeding;
2. infection or other comorbidities;
3. rheumatologic diseases;
4. chronic pain in another joint;
5. chronic use of corticosteroids and immunosuppressants.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-05-08 (Actual); Primary Completion 2016-05-08 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of the research participant after cell transplantation over 12 months | The clinical evaluations will be performed 7 and 15 days and 1, 3, 6 and 12 months after a treatment application
  The function of the temporomadibular joint will be evaluated through the system used for the diagnostic classification "Research Diagnostic Criteria for Temporomandibular Disorders" (RDC/TMD).

SECONDARY OUTCOMES:
Regeneration of articular cartilage after cellular transplantation | The imaging tests (by computed tomography) will be performed 6 and 12 months after the cellular transplantation
  The participant will be submitted to the image examination (computed tomography) for evaluation of the articular osteochondral tissue.
Improvement of the researcher's quality of life after cell transplantation over 12 months | The questionnaires will be applied will be performed 7 and 15 days and 1, 3, 6 and 12 months
  The participants will be evaluated according to the questionnaire "Research Diagnostic Criteria for Temporomandibular Disorders" (RDC/TMD) to evaluate satisfaction with experimental treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Radovan Borojevic, Study Chair — Faculty of Medicine of Petrópolis; Paulo Guimarães, Study Director — Faculty of Medicine of Petrópolis; Ricardo Tesch, Principal Investigator — Faculty of Medicine of Petrópolis
Locations (1):
- Faculdade de Medicina de Petrópolis, Petrópolis, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided